CLINICAL TRIAL: NCT07142460
Title: The Effect of Digital Stories on Nursing Students' Medical Error Tendencies and Safe Parenteral Drug Administration Self-Efficacy
Brief Title: The Effect of Digital Stories on Nursing Students' Medical Error and Safe Drug Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HakimeAslan
Record Dates: First submitted 2025-08-17; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Nursing Students
Keywords: Digital story; Medical error,; Nursing education,; Self-efficacy,; Students
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital story (Experimental)
  Interventions: Behavioral: Intervention
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Intervention — The students in the experimental group were shared the digital stories prepared for drug applications from the WhatsApp group and were asked to watch them for two weeks. Students were able to watch the stories on their mobile phones at the time and frequency they wanted. During 2 weeks, the researchers met with the students twice in the classroom environment and received feedback on the digital stories. Feedbacks about the real meaning of the stories and their contribution to education were obtained by using discussion and question-answer methods. Each student explained their opinions about the stories and had the opportunity to think deeply about them by receiving feedback from their classmates.
  Arms: Digital story

SUMMARY:
Aim This study aimed to determine the effect of digital stories on nursing students' medical error tendencies and safe parenteral drug administration self-efficacy.

Method The study was conducted between May-July 2024 with 64 students (Intervention: 31, Control: 33) studying at the Faculty of Nursing of a university in eastern Turkey and taking the first year nursing principles course. The data were obtained by using 'Personal Information Form', 'Medical Error Tendency Scale, Drug and Transfusion Practices Subscale' and 'Safe Parenteral Drug Administration Self-Efficacy Scale'. During the research process, the students in the experimental group were shared the digital stories prepared for drug applications from the WhatsApp group and were asked to watch them for two weeks.During 2 weeks, the researchers met with the students twice in the classroom environment and received feedback on the digital stories. Students in the control group continued the routine theoretical and practical process.

DETAILED DESCRIPTION:
Digital stories provide personalised learning opportunities that enable students to observe educational environments and events, access them anytime and anywhere, and acquire self-directed learning skills. This method is increasingly being used in education because it offers personalised learning opportunities and enhances teacher-student interaction. In this study, the effects of watching and analysing digital stories prepared for drug administration on nursing students' medical error tendencies and the development of their self-efficacy levels in parenteral drug administration were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or over
* To be enrolled in the first year of nursing,
* To received training on drug administration for the first time,
* To have no physical disabilities related to vision, hearing and motor skills,
* To have a smart mobile phone with Android/IOS operating system,
* To volunteer to participate in the study.

Exclusion Criteria:

* To repeated the first grade
* Not volunteering to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Efeect of Medical Error Tendency | 2 week
  For the pre-test data, 'Individual Introduction Form' and 'Medical Error Tendency Scale' were given to the students and they were asked to fill them in.
  At the end of 2 weeks, the 'Medical Error Tendency Scale' was applied again at the end of the 2nd week to see the change in the medical error tendency levels of the students who were trained with digital stories teaching method for 2 weeks. Medical Error Tendency Scale: It was developed by Özata and Altunkan to measure the medical error tendencies of nurses. The scale consists of 49 items and 5 different sub-dimensions, and the sub-dimension used in this study, the sub-dimension of medication and transfusion practices, consists of 18 items. The higher the mean score of the scale, the lower the tendency of nurses to make medical errors.

SECONDARY OUTCOMES:
Effect of Safe Parenteral Drug Administration Self-Efficacy | 2 weeks
  Safe Parenteral Drug Administration Self-Efficacy Scale: The scale developed to determine the self-efficacy of nurses regarding parenteral drug administration consists of 76 items and one dimension. The scale is a 5-point Likert-type scale and 1: Completely disagree, 2: Disagree, 3: Undecided, 4: Agree, 5: Strongly agree. A minimum score of 76 and a maximum score of 380 can be obtained from the scale. The higher the score obtained from the scale, the higher the self-efficacy of nurses regarding safe parenteral drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Hakime Aslan, Principal Investigator — Faculty of Nursing
Locations (1):
- Inonu University, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No